CLINICAL TRIAL: NCT04651205
Title: Effects of Vitamin B1 and Magnesium Supplements on Glucose Metabolism in Adults Voluntarily Following Reduced-carbohydrate Diets: a Proof of Concept Intervention Study
Brief Title: B1 and Magnesium Supplements on Glucose Metabolism in Low-carb Dieters
Acronym: B-Mag
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Chaitong Churuangsuk, MD, Principal investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200180160
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Diet, Carbohydrate-restricted
Keywords: glucose; low-carbohydrate; magnesium; thiamine; supplement
MeSH Terms: interventions — Thiamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Untreated (No Intervention): This control group will be untreated for 8 weeks as to be a controlled group. Then all participants in the control group will be randomised again to either Mg-B1 or B1-Mg groups for another 8 weeks (delayed-start intervention).
- Mg-B1 early start (Experimental): Participants in the Mg-B1 are the 'early start' group where they will receive 400 mg of Mg per day for 4 weeks then add on 100 mg of B1 per day for another 4 weeks, a total duration of 8 weeks (MgB1).
  Interventions: Dietary Supplement: vitamin B1 and magnesium supplements
- B1-Mg early start (Experimental): Participants in the B1-Mg are the 'early start' group where they will receive 100 mg of B1 per day for 4 weeks then add on 400 mg of Mg per day for another 4 weeks, a total duration of 8 weeks (B1Mg).
  Interventions: Dietary Supplement: vitamin B1 and magnesium supplements

INTERVENTIONS:
Dietary Supplement: vitamin B1 and magnesium supplements — vitamin B1 - 100 mg/day magnesium - 400 mg/day
  Arms: B1-Mg early start; Mg-B1 early start

SUMMARY:
Magnesium (Mg) and thiamine (vitamin B1) are micronutrients involved in the regulation of blood sugar level. Avoidance of wholegrains or fruits and starchy vegetables could impact on Mg and vitamin B1 intakes and status. Although supplementation can be recommended alongside low-carbohydrate high fat diets (LCHF) diets, its benefits have never been studied before.

This study aims to test the effect of Mg and vitamin B1 supplements on glucose metabolism in people following any LCHF diet.

DETAILED DESCRIPTION:
It is clear that Mg involves in both type 2 diabetes (T2D) prevention and management, and following LCHF diets, avoidance of wholegrains, fruits and starchy vegetables, could have a negative impact on Mg and B1 intakes and status. A systematic review of LCHF diets and micronutrients confirmed that Mg and B1 intakes were reduced by 50% and 70% following LCHF diets compared to baseline normal carbohydrate diets, and could be as low as 40% and 75% of recommended intakes for Mg and B1 respectively. Although supplementation can be recommended alongside LCHF diets, not all LCHF dieters take supplements, and their benefits during LCHF diets have never been studied before.

Rationale We hypothesise that people who have been following LCHF diets without taking supplement are potentially at risk of Mg/B1 insufficiency, with negative impact on glucose metabolism.

Objective

1. To investigate potential efficacy of Mg/B1 supplementation on glucose metabolism (mechanistic efficacy/proof of concept) in adults already voluntarily following LCHF
2. To investigate effect of Mg/B1 supplementation on Mg/B1 status in adults already voluntarily following LCHF, who are at risk of Mg/B1 inadequacy
3. To test capabilities of measures, procedures, recruitment criteria, and operational strategies that are under consideration for use in a subsequent, larger, study.
4. To identify barriers to successful study completion
5. To evaluate acceptability of methods and instruments to participants

Study design: This is a mechanistic efficacy/proof of concept, intervention study with a use of a randomised-start design. All participants will be assigned to the same intervention but at different times.

There are 3 groups of the study - 2 interventions and 1 control group:

1. 400 mg of Mg per day for 4 weeks then add on 100 mg of B1 per day for another 4 weeks, a total duration of 8 weeks (MB).
2. 100 mg of B1 per day for 4 weeks then add on 400 mg of Mg per day for another 4 weeks, a total duration of 8 weeks (BM).
3. Untreated: Participants with delayed entry (untreated) for 8 weeks (Con)

Assessment: Baseline, 4 weeks, and 8 weeks after intervention/untreated period

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years and older
2. have been following LCHF diets for at least 2 months
3. carbohydrate intake is less than 130 g/day or less than 26% of energy intake
4. have stable body weight (weight change ≤ 2 kg within two months period)
5. no diagnosed or suspected eating disorder.

Exclusion Criteria:

1. currently taking Mg and B1 supplements within the last 3 months
2. underweight defined by BMI below 18.5 kg/m2
3. have been diagnosed with T1DM or other types of diabetes apart from T2DM.
4. if potential participants have been diagnosed with T2DM, they will be excluded if they are on anti-diabetic drugs and/or insulin (see 7.) or if they are currently following a complete diet for weight loss (e.g. meal replacement, Slimfast, etc.)
5. currently taking anti-diabetic drugs (e.g. metformin, sulfonylurea, GLP-1 agonist, DPP4-inhibitor, SGLT-2 inhibitor, etc) nor insulin use
6. currently taking medications that interact with Mg supplement
7. currently taking medications that may affect glucose metabolism such as steroids, hormonal therapy (e.g. hormone replacement therapy in postmenopausal), antipsychotics.
8. pregnant and lactating women.
9. have gastrointestinal tract diseases e.g. Inflammatory bowel diseases, irritable bowel syndrome, coeliac disease, including other diseases that involve malabsorption.
10. have kidney disease or impair renal function
11. have auto-immune/connective tissue diseases, malignancy.
12. currently dieting or losing 5% of body weight or more during the last 6 months (or planning to do so in the following year).
13. currently participating in other intervention studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
fasting plasma glucose | 8 weeks
  changes from baseline and after supplementation
fasting insulin | 8 weeks
  changes from baseline and after supplementation
homeostatic model assessment of insulin resistance (HOMA-IR) | 8 weeks
  changes from baseline and after supplementation
incremental area under the curve (iAUC) of glucose and insulin after 75 g oral glucose tolerance test | 8 weeks
  changes from baseline and after supplementation
magnesium status | 8 weeks
  changes from baseline and after supplementation
vitamin B1 status | 8 weeks
  changes from baseline and after supplementation

SECONDARY OUTCOMES:
lipid profile: plasma Triglyceride, Total cholesterol, LDL-cholesterol, HDL-cholesterol | 8 weeks
  changes from baseline and after supplementation
plasma hs-CRP | 8 weeks
  changes from baseline and after supplementation
plasma IL-6 | 8 weeks
  changes from baseline and after supplementation
sRAGE | 8 weeks
  changes from baseline and after supplementation
Urine 8-isoprostane | 8 weeks
  , MDA, glycation markers (fructosamine and HbA1c, dermal glycation by skin fluorescence)
plasma 8-isoprostane | 8 weeks
  changes from baseline and after supplementation
plasma fructosamine | 8 weeks
  changes from baseline and after supplementation
HbA1c | 8 weeks
  changes from baseline and after supplementation
dermal glycation by skin fluorescence | 8 weeks
  changes from baseline and after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Chaitong Churuangsuk, MD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Churuangsuk C, Griffiths D, Lean MEJ, Combet E. Impacts of carbohydrate-restricted diets on micronutrient intakes and status: A systematic review. Obes Rev. 2019 Aug;20(8):1132-1147. doi: 10.1111/obr.12857. Epub 2019 Apr 22. PMID 31006978